CLINICAL TRIAL: NCT02047825
Title: Intervention Focused on Lower Limbs and Functionality in Patients With Multiple Sclerosis
Brief Title: Upper Limbs Intervention in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: DF0048UG
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Dexterity; Upper limbs
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): The patients included in this group will receive an intensive intervention based on upper limbs intervention with exercises added to the usual treatment they receive.
  Interventions: Other: Upper limbs intervention
- Control group (Active Comparator): Patients with multiple sclerosis not included in the intensive intervention. They receive the usual treatment of occupational and physical therapy.
  Interventions: Other: Usual treatment

INTERVENTIONS:
Other: Upper limbs intervention — An 8-week intervention with different exercises will be performed. This intervention will focus on upper limbs. The exercises will include plaster of resistance, elastic bands and other exercises.
  Other Names: Exercise program
  Arms: Experimental group
Other: Usual treatment — Occupational therapy and physiotherapy, twice a week, as usual.
  Other Names: Standard treatment
  Arms: Control group

SUMMARY:
Multiple sclerosis is a chronic and highly disabling disorder with considerable social impact and economic consequences. It is caused by damage to the myelin sheath, the protective covering that surrounds nerve cells. Different areas are affected, including manual dexterity, strength, coordination and function. The objective of this study is to evaluate the improvement in these variables in patients with multiple sclerosis after a 8-weeks intervention focused on upper limbs.

DETAILED DESCRIPTION:
The total estimated prevalence rate of multiple sclerosis has been reported to be 83 per 100 000 for the past three decades. It is also higher in northern countries and between females with a male ratio around 2.0. The highest prevalence rates have been estimated for the age group 35-64 years. The estimated European mean annual Multiple Sclerosis incidence rate is 4.3 cases per 100 000.

Multiple sclerosis can cause a variety of symptoms: hypoesthesia, muscle weakness, abnormal muscle spasms, or difficulty moving; difficulties with coordination and balance; dysarthria, dysphagia, visual problems fatigue and acute or chronic pain syndromes, bladder and bowel difficulties,cognitive impairment, or emotional symptomatology. The investigators focus on the benefits of an intervention on dexterity, strength, coordination and functionality.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple sclerosis.
* Subjects who can complete the assessment battery of tests at the beginning and at the end of the study

Exclusion Criteria:

* Auditive and visual disturbances.
* Cognitive problems.
* Psychiatric pathology.
* Sensorial disturbances.
* Traumatic pathology of the hand.
* Concomitant neurological conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in manual dexterity | baseline, 8 weeks
  Changes from baseline to postintervention in manual dexterity assessed by the Purdue Pegboard test and coin rotation task. The Purdue pegboard test is a timed physical test used to measure manual dexterity. Test subjects are asked to place small pins into holes in the pegboard using a specific hand and following a specific process. The coin rotation task consists of rotate the coin during 10 seconds.

SECONDARY OUTCOMES:
Changes in apraxia | baseline, 8 weeks
  Changes in apraxia from baseline to postintervention is going to be measured using the Apraxia Screen of Tulia. This is a screening test of upper limbs apraxia.
Changes in grip strength | baseline, 8 weeks
  The changes in the grip strength will be measured using a Jamar dynamometer with a standard protocol allowing three attempts on each side. During each measurement, patients were sitting with their shoulder adducted and elbow flexed to 90°. The maximum value achieved from all six attempts was used in analyses. kg/cm2.
Change in fatigue | baseline, 8 weeks
  The fatigue change is going to be measured using the Fatigue Severity Scale, a 9-item scale focus on the severity of fatigue and how much it affects the person's activities and lifestyle in the patients.
Upper limb functioning | baseline, 8 weeks
  The upper limb functioning is going to be measured with the Action Research Arm Test, it is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement).
Pinch strength | baseline, 8 weeks
  Pinch strength is going to be measured using a pinch dynamometer. The participants were asked to perform three repetitions on each side with five seconds rest provided between the measures. This was performed using the alternating-hands method, which allows rest between repetitions as the examiner records information and provides instructions for the alternate hand. Three pinchs were evaluated: lateral, distal and tripod pinch
Tapping speed | baseline, 8 weeks
  The tapping speed will be measured with the finger tapping test.

OTHER OUTCOMES:
Quality of life | Baseline, 8 weeks
  Quality of life is going to be measured using a self-reported questionnaire, the short-form Health Survey, SF-36
Goals achievement | baseline, 8 weeks
  The achievement of the goals of the intervention will be measured with the Goal Attainment Scale, a method of scoring the extent to which patient's individual goals are achieved in the course of intervention.
Functionality | baseline, 8 weeks
  Functionality will be measured with the Functional Independence Measure, a questionnaire. This is the most widely accepted functional assessment measure in use in the rehabilitation community

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ortiz-Rubio A, Cabrera-Martos I, Rodriguez-Torres J, Fajardo-Contreras W, Diaz-Pelegrina A, Valenza MC. Effects of a Home-Based Upper Limb Training Program in Patients With Multiple Sclerosis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Dec;97(12):2027-2033. doi: 10.1016/j.apmr.2016.05.018. Epub 2016 Jun 22. PMID 27343343